CLINICAL TRIAL: NCT00730327
Title: Safety and Effectiveness of the BioEnterics® Intragastric Balloon (BIB®) System to Assist in the Weight Management of Obese Subjects
Brief Title: A Study of BioEnterics® Intragastric Balloon (BIB®) System to Assist in the Weight Management of Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apollo Endosurgery, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IB-005
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIB® (Experimental): Receives BioEnterics® Intragastric Balloon Intervention as well as diet and exercise counseling with the Behavioral Modification Intervention.
  Interventions: Device: BioEnterics® Intragastric Balloon; Other: Behavioral modification
- Control (Other): Control arm receives the Behavioral modification intervention only.
  Interventions: Other: Behavioral modification

INTERVENTIONS:
Device: BioEnterics® Intragastric Balloon — Inflatable balloon inserted into the stomach.
  Other Names: BIB®
  Arms: BIB®
Other: Behavioral modification — Low-calorie diet, food/exercise diary, eating plan, emphasis on exercise

SUMMARY:
Safety and effectiveness of the BIB® System in conjunction with a behavior modification program compared to the behavior modification program alone for weight loss in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI ≥ 30 and ≤ 40;
* Be male or female, between 18 and 65 years of age, inclusive;
* Have a history of obesity (BMI ≥ 30 kg/m2) for at least 2 years and have failed more conservative weight-reduction alternatives, such as supervised diet, exercise and behavioral modification programs;
* Be willing to commit to a long-term low calorie (1000-1500 calories/day) supervised diet;
* Have reasonable weight loss expectations (accept a goal of losing up to 15% of body weight after 26 weeks);
* Be able to follow requirements outlined in the protocol, including complying with the visit schedule and behavioral modification program, and willing to undergo protocol-specific procedures, e.g., endoscopy, local sedation, general anesthesia, upper gastrointestinal radiography (UGI), electrocardiography (EKG), gastric motility testing, and/or clinical laboratory testing;
* Must be willing to take prescribed proton pump inhibitors (PPIs)and other medications as prescribed by the investigator;
* Be able to provide written informed consent and authorization for use and release of Health and Research Study Information;
* Be willing to use contraception (e.g., birth control pills, condoms, abstinence) and avoid pregnancy during the study if female of child-bearing potential.

Exclusion Criteria:

* Any surgery of the foregut excluding uncomplicated cholecystectomy
* History or symptoms of gastrointestinal (GI) surgery (excluding uncomplicated appendectomy), GI obstruction, adhesive peritonitis, and/or hiatal hernia (>/= 2 cm);
* A patulous pyloric channel;
* History or symptoms of esophageal or GI motility disorders (not just those with <40%) as these patients are particularly susceptible to the development of esophagitis;
* History or previous symptoms of delayed Gastric Emptying (GE) and/or delayed GE having been documented on a previously performed gastric scintigraphy study or another previously performed diagnostic study such as a UGI x-ray series;
* Current symptoms of delayed GE;
* A history of myocardial infarction in the previous 6 months: New York Heart Associate (NYHA) Class III or IV (heart failure) or cardiac arrhythmia (e.g., atrial fibrillation);
* Anemia defined as a hemoglobin value for females of <11.3 g/dl and for males < 13.0 g/dl;
* History or symptoms of varices, bowel obstruction, congenital or acquired GI anomalies (e.g., atresias, stenosis, stricture, and/or diverticula), severe renal, hepatic, and/or pulmonary disease;
* History or symptoms of inflammatory bowel disease, such as Crohn's disease or Ulcerative Colitis;
* History or symptoms of uncontrolled or unstable thyroid disease;
* Subjects with a positive test for Helicobacter pylori (H.p.) at screening; subjects may participate in the study if, prior to randomization, they are treated with a pharmacological regimen designed to eradicate their H.p. and subsequently have a negative H.p. breath test indicating that the H.p. has been eradicated
* History or symptoms in the past 24 months of significant irritable bowel syndrome, peritonitis, active esophagitis, gastritis and/or duodenitis, gastric or duodenal ulceration, GI hemorrhage, or GI bleeding;
* Type I diabetes;
* Placement of previous intragastric balloon or similar device;
* Ongoing treatment with anticoagulants, steroids, aspirin, non-steroidal anti-inflammatory drugs (NSAIDS), or other medications known to be gastroduodenal mucosal irritants or to reduce GI motility, and/or an unwillingness to discontinue the use of these concomitant medications;
* Concomitant use of prescription, non-prescription, or over-the-counter weight loss medications or supplements at any time during the study;
* Evidence of untreated psychiatric or eating disorders, such as major depression, schizophrenia, substance abuse, binge eating disorder, or bulimia;
* Pregnancy, breast feeding, or intention of becoming pregnant during the study (if female of childbearing potential;
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study;
* Poor general health, presence of a specific condition, or is in a situation, which in the Evaluating and/or Placing Investigator's opinion may put the subject at significant risk, may confound the study results, may increase the risks associated with endoscopy and/or placement of the BIB, or may interfere significantly with the subject's participation in the study (e.g., HIV, Hepatitis C, or cancer history within the last 5 years)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2008-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Eaton, RN, BSN, Study Director — Apollo Endosurgery, Inc.
Locations (1):
- Apollo Endosurgery, Austin, Texas, United States

REFERENCES:
- [Derived] Gomez V, Woodman G, Abu Dayyeh BK. Delayed gastric emptying as a proposed mechanism of action during intragastric balloon therapy: Results of a prospective study. Obesity (Silver Spring). 2016 Sep;24(9):1849-53. doi: 10.1002/oby.21555. Epub 2016 Jul 28. PMID 27465076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 15 investigational sites across the US, between 6/20/2008 and 10/10/2010. Patients were either enrolled as run-in subjects (mentored cases which were enrolled prior to randomized subjects in order for physicians to gain experience with placing and removing the device) or as subjects for randomization.
Pre-assignment Details: 448 subjects were enrolled (defined as signing the informed consent), 44 of which were run-in subjects. Prior to randomization, 131 subjects were screen failures. 273 subjects were randomized to the BIB (137) and control groups (136). 12 BIB and 6 control subjects discontinued prior to treatment. 125 BIB and 130 control subjects began treatment.
Period: Overall Study
Arm/Group | BIB® | Control
Started | 125 (Started is defined as subjects that began treatment.) | 130
Completed Week 26 | 125 (Week 26 was halfway through the study, at which point the BIB group had their balloon removed.) | 99
Completed | 98 (Completed defined as subjects who completed the Week 52 follow-up visit.) | 93
Not Completed | 27 | 37
Not completed — Lost to Follow-up | 14 | 16
Not completed — Adverse Event | 8 | 1
Not completed — Withdrawal by Subject | 3 | 13
Not completed — Subject withdrew (reason not specified) | 2 | 7

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consisted of the Intent-to-Treat (ITT) population. All baseline characteristics were calculated at the screening visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | BIB® | Control | Total
Number analyzed (Participants) | 125 | 130 | 255
Age, Customized [Number; unit: participants]
  18-19 years | 1 | 0 | 1
  20-29 years | 21 | 18 | 39
  30-39 years | 49 | 37 | 86
  40-49 years | 31 | 54 | 85
  50-59 years | 22 | 16 | 38
  60 years & over | 1 | 5 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 117 | 229
  Male | 13 | 13 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 101 | 106 | 207
  Hispanic | 9 | 7 | 16
  Black (not of Hispanic origin) | 14 | 15 | 29
  Asian | 0 | 0 | 0
  Other | 1 | 2 | 3
BMI [Number; unit: participants] — Subject BMI (kg/m²) was calculated using their baseline weight at screening. Subjects with BMI<30 or >40 were major protocol deviations
  participants
    BMI <30 | 2 | 1 | 3
    BMI ≥30 and <35 | 63 | 57 | 120
    BMI ≥35 and ≤40 | 56 | 70 | 126
    BMI >40 | 4 | 2 | 6
Number of Years Obese [Number; unit: participants]
  < 5 years obese | 20 | 22 | 42
  5-9 years obese | 35 | 26 | 61
  10-19 years obese | 38 | 51 | 89
  20-29 years obese | 18 | 19 | 37
  30-39 years obese | 10 | 6 | 16
  40-49 years obese | 1 | 4 | 5
  50 years obese & over | 0 | 0 | 0
  Unknown | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Excess Weight Loss (%EWL)
Description: The first co-primary effectiveness measure, was mean percent excess weight loss (% EWL) at 9 months (3 months after the balloon was removed for the BIB group). Percent EWL was calculated using the 1983 Met Life tables for determination of ideal body weight, per the protocol-defined primary effectiveness endpoint.
  Percent EWL was calculated as %EWL= (weight loss divided by excess weight)*100, where Weight loss = Baseline weight - selected follow-up weight, and Excess weight = Baseline weight - ideal weight.
Time Frame: 9 months
Population: Randomized participants in the intent-to-treat (ITT) population who completed the 39 week (month 9) follow-up visit (with last observed carried forward).
Measure: Mean (Standard Deviation); unit: percentage of EWL
Arm/Group | BIB® | Control
Number analyzed (Participants) | 91 | 95
percentage of EWL | 26.52 (20.70) | 9.67 (15.11)

2. Primary Outcome: Percentage of BIB Treated Participants With Significantly Greater Weight Loss Than the Control Group
Description: The second co-primary effectiveness measure was the percentage of BIB treated participants with significantly greater weight loss than the control group at 9 months. Significantly greater weight loss was defined as ≥ 15% EWL over the mean %EWL of the control group.
  %EWL= (weight loss divided by excess weight) * 100, where Weight loss = Baseline weight - selected follow-up weight and Excess weight = Baseline weight - ideal weight.
  Ideal weight was determined by using the 1983 Metropolitan Life Height and Weight Table.
Time Frame: 9 months
Population: Randomized participants in the ITT population who completed the 39 week (9 month) follow-up visit (with last observation carried forward).
Measure: Number (95% Confidence Interval); unit: percentage of BIB participants
Arm/Group | BIB®
Number analyzed (Participants) | 91
percentage of BIB participants
  15% EWL over the control group mean | 45.60 [36.67 to 54.75]
  25% EWL over the control group mean | 32.8 [24.67 to 41.77]

3. Secondary Outcome: Percent of Participants With Comorbid Conditions
Description: The percent of participants with a comorbid condition (type 2 diabetes, hypertension, or dyslipidemia) at Week 26 (6 months, balloon removal for BIB group), Week 39 (9 months), and Week 52 (12 months) as compared to baseline.
  Comorbid conditions were measured and diagnosed by lab tests and vital signs. Type 2 Diabetes was diagnosed if participants' had a Fasting Plasma Glucose (FPG) ≥126 mg/dL, or symptoms of diabetes plus casual plasma glucose concentration ≥200 mg/dL.
  Hypertension was diagnosed if participants' blood pressure measured ≥140 mmHg systolic or ≥90 mmHg diastolic.
  Dyslipidemia was diagnosed if participants' labs measured: LDL ≥160 mg/dL, Total Cholesterol ≥240 mg/dL, Serum Triglycerides ≥200 mg/DL, HDL <50 mg/dL (male) or <40 mg/dL (female).
Time Frame: Baseline, Week 26, Week 39, Week 52
Population: Randomized participants in the ITT population that provided data at that timepoint. n=number of participants who provided lab data at that visit (number of participants varied as not all participants provided all lab data at each visit).
Measure: Number; unit: percentage of participants
Arm/Group | BIB® | Control
Number analyzed (Participants) | 125 | 130
percentage of participants
  Diabetes-Baseline (BIB n=124, Control n=130) | 7.3 | 6.2
  Diabetes-Week 26 (BIB n=100, Control n=94) | 3.0 | 4.3
  Diabetes-Week 39 (BIB n=102, Control n=94) | 4.9 | 3.2
  Diabetes-Week 52 (BIB n=95, Control n=94) | 3.2 | 5.3
  Hypertension-Baseline (BIB n=125, Control n=130) | 26.4 | 28.5
  Hypertension-Week 26 (BIB n=124, Control n=91) | 17.7 | 19.8
  Hypertension-Week 39 (BIB n=91, Control n=95) | 15.4 | 21.1
  Hypertension-Week 52 (BIB n=98, Control n=92) | 11.2 | 22.8
  Dyslipidemia-Baseline (BIB n=125, Control n=130) | 39.2 | 30.0
  Dyslipidemia-Week 26 (BIB n=102, Control n=94) | 31.4 | 27.7
  Dyslipidemia-Week 39 (BIB n=102, Control n=95) | 28.4 | 28.4
  Dyslipidemia-Week 52 (BIB n=96, Control n=94) | 30.2 | 26.6

4. Secondary Outcome: Change in Quality of Life (SF-36)
Description: The change in quality of life from baseline to 9 months was measured by the Short Form 36 (SF-36) questionnaire. The SF-36 health survey consists of 36 questions that evaluate 8 discrete domains: Physical Functioning (Physical Func), Social Functioning (Social Func), Bodily Pain, General Health Perceptions (General Health), Vitality, Role limitations due to emotional problems (Role-Emotional), Role limitations due to physical health (Role Physical), and Mental Health. The score for each domain ranges from 0 (poorest health status) to 100 (best health status). The BIB group's mean scores for each SF-36 domain at baseline and week 39 were compared to the control group's mean scores.
Time Frame: Baseline, Week 39
Population: Randomized participants in the ITT population that provided data at each timepoint. n = number of participants (number of participants varied as not all participants provided data on all questionnaire items at both timepoints).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIB® | Control
Number analyzed (Participants) | 123 | 130
units on a scale
  Physical Func-Baseline (BIB n=122, Control n=130) | 71.4 (22.09) | 73.7 (21.14)
  Physical Func-Week 39 (BIB n=98, Control n=92) | 90.0 (14.26) | 85.4 (15.5)
  Role Physical-Baseline (BIB n=123, Control n=130) | 78.5 (21.59) | 80.3 (23.07)
  Role Physical-Week 39 (BIB n=98, Control n=93) | 93.0 (13.56) | 85.6 (20.89)
  Bodily Pain-Baseline (BIB n=123, Control n=130) | 72.8 (21.88) | 75.4 (22.34)
  Bodily Pain-Week 39 (BIB n=99, Control n=93) | 84.9 (18.84) | 76.2 (23.91)
  General Health-Baseline (BIB n=123, Control n=128) | 61.9 (20.22) | 63.4 (20.11)
  General Health-Week 39 (BIB n=99, Control n=93) | 79.1 (16.53) | 68.6 (20.67)
  Vitality-Baseline (BIB n=123, Control n=130) | 52.7 (18.19) | 53.0 (19.11)
  Vitality-Week 39 (BIB n=99, Control n=93) | 67.6 (17.74) | 58.3 (21.08)
  Social Func-Baseline (BIB n=123, Control n=130) | 80.5 (21.89) | 80.8 (23.30)
  Social Func-Week 39 (BIB n=99, Control n=93) | 92.6 (13.35) | 83.3 (22.14)
  Role Emotional-Baseline (BIB n=123, Control n=130) | 84.0 (22.65) | 84.6 (20.81)
  Role Emotional-Week 39 (BIB n=98, Control n=93) | 92.2 (15.55) | 86.8 (19.75)
  Mental Health-Baseline (BIB n=123, Control n=130) | 74.0 (17.91) | 73.7 (16.60)
  Mental Health-Week 39 (BIB n=99, Control n=93) | 80.1 (15.82) | 72.5 (18.09)

5. Secondary Outcome: Change in Quality of Life (IWQOL-Lite)
Description: The change in quality of life from baseline to 12 months was measured by the Impact of Weight on Quality of Life - Lite (IWQOL-Lite) questionnaire. IWQOL-Lite consists of 31 scale items to assess obesity-related quality of life, and total score ranges from 0 (worst) to 100 (best). The BIB group's mean IWQOL-Lite score at baseline, Week 26 (6 months, balloon removal for BIB group), Week 39 (9 months) and Week 52 (12 months) were compared to the control group's mean scores at the same timepoints.
Time Frame: Baseline, Week 26, Week 39, Week 52
Population: Randomized participants in the ITT population that provided data at each timepoint. n = number of participants (number of participants varied as not all participants provided data on questionnaire at both timepoints).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIB® | Control
Number analyzed (Participants) | 121 | 127
units on a scale
  Baseline (BIB n=121, Control n=127) | 68.40 (18.733) | 68.55 (17.356)
  Week 26 (BIB n=103, Control n=94) | 84.64 (12.888) | 76.67 (16.472)
  Week 39 (BIB n=99, Control n=93) | 85.78 (14.411) | 78.58 (16.833)
  Week 52 (BIB n=97, Control n=94) | 85.79 (15.424) | 79.85 (16.189)

6. Secondary Outcome: Change in Participant Depression (Beck Depression Inventory II)
Description: Participants were assessed for depression using the Beck Depression Inventory II (BDI-II) questionnaire. The BDI-II consists of 21 questions to measure depressive symptoms and severity. The overall score ranges from 0-63, where higher total scores indicate more severe depressive symptoms. A total score of 0-13 is considered a minimal range, 14-19 is mild, 20-28 is moderate and 29-63 is interpreted as severe depressive symptoms. The mean BDI-II score for the BIB and control groups were assessed at baseline and at key timepoints: Week 26 (month 6, balloon removal for BIB group), Week 39 (month 9), and Week 52 (month 12, study completion).
Time Frame: Baseline, Week 26, Week 39, Week 52
Population: Randomized participants in the ITT population that provided data at each visit. n=the number of participants (number of participants varies as not all participants completed the questionnaire at each visit)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIB® | Control
Number analyzed (Participants) | 124 | 130
units on a scale
  Baseline (BIB n=124, Control n=130) | 7.7 (7.92) | 8.4 (7.79)
  Week 26 (BIB n=104, Control n=95) | 3.7 (4.83) | 7.0 (8.30)
  Week 39 (BIB n=99, Control n=93) | 3.6 (5.12) | 6.3 (6.68)
  Week 52 (BIB n=97, Control n=95) | 3.9 (6.42) | 5.7 (7.30)

7. Post Hoc Outcome: Change in BMI
Description: Post-Hoc effectiveness analyses were performed per the request of FDA after the study closed, therefore the protocol was not amended. The data was analyzed to determine the change in participant's Body Mass Index (BMI) at key timepoints throughout the study. The mean BMI for the BIB and Control group was assessed at baseline, Week 26 (6 months, balloon removal for BIB group), Week 39 (9 months), and Week 52 (12, months, study completion).
Time Frame: Baseline, Week 26, Week 39, Week 52
Population: Randomized participants in the ITT population who provided weight data at that visit. n=number of participants (number of participants varies as not all participants provided data at each timepoint).
Measure: Mean (Standard Deviation); unit: kg/m²
Arm/Group | BIB® | Control
Number analyzed (Participants) | 125 | 130
kg/m²
  Baseline (BIB n=125, Control n=130) | 35.20 (3.165) | 35.43 (2.650)
  Week 26 (BIB n=117, Control n=91) | 31.43 (3.762) | 33.61 (3.253)
  Week 39 (BIB n=91, Control n=95) | 31.85 (4.035) | 33.83 (3.300)
  Week 52 (BIB n=98, Control n=92) | 32.50 (4.177) | 33.96 (3.517)

8. Post Hoc Outcome: Percent EWL (Using BMI=25 kg/m²)
Description: Post-Hoc effectiveness analyses were performed per the request of FDA after the study closed, therefore the protocol was not amended. The data was analyzed to determine participants' mean %EWL (using a BMI=25 kg/m² as ideal weight) at key timepoints. Participants' mean %EWL was assessed at Week 26 (6 months, balloon removal for BIB group), Week 39 (9 months), and Week 52 (12, months, study completion).
  Percent EWL was calculated as %EWL= (weight loss divided by excess weight)*100, where Weight loss = Baseline weight - selected follow-up weight, and Excess weight = Baseline weight - ideal weight, where ideal weight was BMI=25.
Time Frame: Baseline, Week 26, Week 39, Week 52
Population: Randomized participants in the ITT population with last observed carried forward (number of participants varies as not all participants provided data at each timepoint)
Measure: Mean (Standard Deviation); unit: percentage of EWL
Arm/Group | BIB® | Control
Number analyzed (Participants) | 125 | 130
percentage of EWL
  Week 26 (BIB n=117, Control n=91) | 38.4 (27.61) | 12.1 (18.58)
  Week 39 (BIB n=91, Control n=95) | 34.6 (28.4) | 12.3 (19.33)
  Week 52 (BIB n=98, Control n=92) | 29.0 (30.70) | 11.1 (20.67)

9. Post Hoc Outcome: Percent Total Body Weight Loss (%TBWL)
Description: Post-Hoc effectiveness analyses were performed per the request of FDA after the study closed, therefore the protocol was not amended. The data was analyzed to determine participants' Percent Total Body Weight Loss (%TBWL) at key timepoints throughout the study. The mean %TBWL for the BIB and Control group was assessed at baseline, Week 26 (6 months, balloon removal for BIB group), Week 39 (9 months), and Week 52 (12, months, study completion).
Time Frame: Baseline, Week 26, Week 39, Week 52
Population: Randomized participants in the ITT population with last observation carried forward. n=number of participants (number of participants varies as not all participants provided data at each timepoint).
Measure: Mean (95% Confidence Interval); unit: percentage of TBWL
Arm/Group | BIB® | Control
Number analyzed (Participants) | 125 | 130
percentage of TBWL
  Week 26 (BIB n=117, Control n=91) | 10.2 [9.0 to 11.4] | 3.3 [2.4 to 4.2]
  Week 39 (BIB n=91, Control n=93)5 | 9.1 [7.9 to 10.3] | 3.4 [2.4 to 4.3]
  Week 52 (BIB n=98, Control n=92) | 7.6 [6.2 to 8.9] | 3.1 [2.0 to 4.1]

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data was collected over a period of 12 months.
Description: AE data was collected beginning with the start of treatment (BIB placement and behavioral modification program for BIB group; behavioral modification program alone for the Control group) and at follow-up visits throughout the study, for a total of 12 months. Both device-related and non-device-related AEs are reported below.
Groups:
- Control: Control arm receives the Behavioral modification intervention only. Behavioral modification: Low-calorie diet, food/exercise diary, eating plan, emphasis on exercise
Arm/Group | BIB® | Control
Serious Adverse Events (participants affected / at risk) | 19/125 | 8/130
Other Adverse Events (participants affected / at risk) | 124/125 | 92/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIB® (N=125) | Control (N=130)
Chronic myelogenous leukemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Event determined to be not-device related for BIB group.
Syncope (Cardiac disorders) | 1 (1) | 0 (0) — Event determined to be not-device related for BIB group.
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0) — Event determined to be not-device related for BIB group.
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) — Event determined to be not-device related for BIB group.
Ventral hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) — Event determined to be not-device related for BIB group.
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Event determined to be not-device related for BIB group.
Device Intolerance (Investigations) | 8 (8) | 0 (0)
Gastric outlet obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Defective device (General disorders) | 1 (1) | 0 (0) — Abdominal cramping due to defective device (bacterial overgrowth).
Choledocholithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) — Event determined to be not-device related for BIB group.
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Giardia lamblia infection (Infections and infestations) | 1 (1) | 0 (0) — Event determined to be not-device related for BIB group.
Viral gastroparesis (Infections and infestations) | 1 (1) | 0 (0) — Event determined to be not-device related for BIB group.
Osteoarthritis of the hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Event determined to be not-device related for BIB group.
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Event determined to be not-device related for BIB group.
Breast abscess (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Event determined to be not-device related for BIB group.
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1) — Event determined to be not-device related for BIB group.
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Laryngospasm during BIB placement (procedure-related)
Hemithyroidectomy (Endocrine disorders) | 0 (0) | 1 (1)
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Motor vehicle accident with nasal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Herniated lumbar disc (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Renal cell carcinoma with nephrectomy (Renal and urinary disorders) | 0 (0) | 1 (1)
Bilateral vertebral artery hypoplasia (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIB® (N=125) | Control (N=130)
Abdominal Distension (Gastrointestinal disorders) | 23 (23) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 81 (81) | 5 (5)
Abdominal Pain Upper (Gastrointestinal disorders) | 23 (23) | 0 (0)
Constipation (Gastrointestinal disorders) | 31 (31) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 25 (25) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 30 (30) | 0 (0)
Eructation (Gastrointestinal disorders) | 29 (29) | 0 (0)
Flatulence (Gastrointestinal disorders) | 14 (14) | 0 (0)
Gastroesophageal Reflux Disease (GERD) (Gastrointestinal disorders) | 38 (38) | 6 (6)
Impaired Gastric Emptying (Gastrointestinal disorders) | 16 (16) | 5 (5)
Nausea (Gastrointestinal disorders) | 112 (112) | 7 (7)
Vomiting (Gastrointestinal disorders) | 97 (97) | 7 (7)
Asthenia (General disorders) | 10 (10) | 0 (0)
Fatigue (General disorders) | 9 (9) | 0 (0)
Bronchitis (Infections and infestations) | 9 (9) | 11 (11)
Ear Infection (Infections and infestations) | 5 (5) | 4 (4)
Nasopharyngitis (Infections and infestations) | 6 (6) | 7 (7)
Pharyngitis streptococcal (Infections and infestations) | 4 (4) | 6 (6)
Sinusitis (Infections and infestations) | 11 (11) | 19 (19)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 13 (13)
Viral infection (Infections and infestations) | 6 (6) | 0 (0)
Medical device complication (Injury, poisoning and procedural complications) | 8 (8) | 0 (0)
Post procedural pain (Injury, poisoning and procedural complications) | 9 (9) | 0 (0)
Blood cholesterol increased (Investigations) | 6 (6) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 17 (17) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Headache (Nervous system disorders) | 11 (11) | 7 (7)
Anxiety (Psychiatric disorders) | 5 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 6 (6)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 4 (4)
Vitamin B1 decreased (Investigations) | 0 (0) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Migraine (Nervous system disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No